CLINICAL TRIAL: NCT03733925
Title: A Phase-IV, Multicenter, Noncomparative, Open-Label Study Evaluating the Safety and Efficacy of Golimumab (a Fully Human Anti-TNFα Monoclonal Antibody, Administered Subcutaneously) in the Treatment of Indian Patients With Active Spondyloarthropathy of Ankylosing Spondylitis or Psoriatic Arthritis
Brief Title: A Study of Golimumab in the Treatment of Indian Participants With Active Spondyloarthropathy of Ankylosing Spondylitis or Psoriatic Arthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Private Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108559; CNTO148SPD4001 (Other: Johnson & Johnson Private Limited)
Record Dates: First submitted 2018-11-05; First posted 2018-11-07 (Actual); Results first posted 2023-01-20 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Spondylitis, Ankylosing; Arthritis, Psoriatic
MeSH Terms: conditions — Spondylitis, Ankylosing; Arthritis, Psoriatic | interventions — golimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Golimumab (Experimental): Participants will receive golimumab 50 milligram (mg) subcutaneous (SC) injection at Week 0 and every 4 weeks (q4w) thereafter through Week 24. Concomitant medications may be allowed on a case by case basis as per the physician's judgement.
  Interventions: Drug: Golimumab

INTERVENTIONS:
Drug: Golimumab — Participants will receive golimumab 50 mg SC injections at Week 0 and q4w thereafter through Week 24.
  Other Names: SIMPONI

SUMMARY:
The purpose of this study is to assess the safety of subcutaneous (SC) golimumab in participants with active Ankylosing Spondylitis (AS) or Psoriatic Arthritis (PsA) over 24 weeks.

DETAILED DESCRIPTION:
This post-marketing study will evaluate safety and efficacy profile of golimumab (a fully human anti-Tumour Necrosis Factor alpha [TNF-alpha] monoclonal antibodies [mAb], administered subcutaneously) in a real-world in Indian participants with active spondyloarthropathy of ankylosing spondylitis (AS) or psoriatic arthritis (PsA). AS is a chronic inflammatory disease of unknown etiology that involves the sacroiliac joints, axial skeleton, entheses, and peripheral joints. PsA is a chronic, inflammatory, usually rheumatoid factor negative arthritis that is associated with psoriasis. Golimumab binds with high affinity to human TNF-alpha and inhibits TNF-alpha bioactivity, TNF-alpha-mediated cell cytotoxicity and TNF-alpha mediated endothelial cell activation. Golimumab also induces activation of complement-mediated cell lysis and reduces the development of arthritis. Study evaluation includes efficacy (efficacy parameters for AS and PsA) and safety. Participant's safety will be monitored throughout the study. The total duration of study will be approximately 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

For participants with Ankylosing Spondylitis (AS):

* Have a diagnosis of definite AS (according to the Modified New York Criteria)
* Either has an inadequate response (defined as Bath Ankylosing Spondylitis Disease Activity Index [BASDAI] greater than or equal to [>=]4) to current or past therapies (including biologics naïve participants). Participants who were receiving non-steroidal anti-inflammatory drugs (NSAIDs) or disease-modifying antirheumatic drugs (DMARDs) had to have received continuous therapy for 3 months at the highest recommended doses or had to have been unable to receive a full 3-month course of full-dose NSAID or DMARD therapy because of intolerance, toxicity, or contraindications. Maximum recommended dosages for DMARDs if used, would be: methotrexate 25 milligram per week (mg/week), oral corticosteroids (less than or equal to [<=]10 milligram per day [mg/day] of prednisone or equivalent) or sulfasalazine 3 gram per day (g/day)

For participants with Psoriatic Arthritis (PsA):

* Have PsA that was diagnosed at least 6 months prior to the first administration of study drug (according to the ClASsification criteria for Psoriatic ARthritis [CASPAR])
* Have at least 1 of the PsA subsets: Distal Interphalangeal (DIP) joint arthritis, polyarticular arthritis with the absence of rheumatoid nodules, arthritis mutilans, asymmetric peripheral arthritis, or spondylitis with peripheral arthritis
* Are negative for rheumatoid factors according to the reference range of the local laboratory conducting the test

Exclusion Criteria:

* Are pregnant, nursing, or planning a pregnancy or fathering a child during the study or within 6 months after receiving the last administration of study drug
* Have a known hypersensitivity to human immunoglobulin proteins or other components of golimumab
* Have a history of latent or active granulomatous infection, including histoplasmosis, or coccidioidomycosis, prior to screening
* Have a chest radiograph within 3 months prior to the first administration of study drug that shows an abnormality suggestive of a malignancy or current active infection, including tuberculosis (TB)
* Have had a nontuberculous mycobacterial infection or opportunistic infection (for example, cytomegalovirus, pneumocystosis, aspergillosis) within 6 months prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Private Limited Clinical Trial, Study Director — Johnson & Johnson Private Limited
Locations (9):
- India (9):
  - ChanRe Rheumatology And Immunology Center And Research, Bangalore
  - Apollo Hospitals, Bhubaneswar
  - Chennai Meenakshi Multispeciality Hospital, Chennai
  - Nizams Institute of Medical Sciences NIMS, Hyderabad
  - Apollo Multispeciality Hospital Ltd, Kolkata
  - All India Institute of Medical Sciences, New Delhi
  - Sir Ganga Ram Hospital, New Delhi
  - Indraprastha Apollo Hospital, New Delhi
  - Sancheti Institute for Orthopedics & Rehabilitation, Pune

RESULTS

PARTICIPANT FLOW:
Groups:
- Golimumab (Simponi): Participants with active spondyloarthropathy of AS or PsA received golimumab 50 milligrams (mg) subcutaneous (SC) injection at Week 0 and every 4 weeks (q4w) thereafter through Week 24.
Period: Overall Study
Arm/Group | Golimumab (Simponi)
Started | 100
Participants With Psoriatic Arthritis (PsA) | 50
Participants With Ankylosing Spondylitis (AS) | 50
Completed | 94
Not Completed | 6
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 2
Not completed — Adverse Event | 2
Not completed — Non-Compliance with Study Drug | 1

BASELINE CHARACTERISTICS:
Arm/Group | Golimumab (Simponi)
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.7 (12.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 78
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Indian | 100
Region of Enrollment [Count of Participants; unit: Participants]
  India | 100

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product which does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to that medicinal product. Any AE that occurred at or after the initial administration of study drug through the day of last dose plus 8 weeks was considered to be TEAE.
Time Frame: Up to Week 32
Population: Safety analysis set (SAS) included all participants who were enrolled and received at least one dose of the study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Golimumab (Simponi)
Number analyzed (Participants) | 100
Participants
  Ankylosing Spondylitis (AS): number analyzed (Participants) | 50
  Ankylosing Spondylitis (AS) | 10
  Psoriatic Arthritis (PsA): number analyzed (Participants) | 50
  Psoriatic Arthritis (PsA) | 18

2. Primary Outcome: Number of Participants With Treatment Emergent Serious Adverse Events (SAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product which does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to that medicinal product. SAE was any untoward medical occurrence that at any dose may result in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product. Any AE that occurred at or after the initial administration of study drug through the day of last dose plus 8 weeks was considered to be TEAE.
Time Frame: Up to Week 32
Population: SAS included all participants who were enrolled and received at least one dose of the study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Golimumab (Simponi)
Number analyzed (Participants) | 100
Participants
  AS: number analyzed (Participants) | 50
  AS | 2
  PsA: number analyzed (Participants) | 50
  PsA | 2

3. Secondary Outcome: Percentage of Ankylosing Spondylitis (AS) Participants With at Least 20 Percent (%) Improvement in the Assessment of SpondyloArthritis International Society (ASAS20) Criteria at Week 14
Description: ASAS 20 response criteria was defined as an improvement from baseline of greater than (>)20% and >1 unit in at least 3 of following 4 ASAS domains on scale of 0-10 units and no worsening from baseline of >20% and >1 unit in the remaining ASAS domain on a scale of 0-10 units. The 4 ASAS domains were as follows (0-10 units numerical rating scale [NRS]): Patient's global assessment (PGA) of disease:0=not active spondylitis, 10=very active spondylitis; total and night Spinal pain: 0=no pain, 10=most severe pain; bath ankylosing spondylitis functional index (BASFI, self-assessment of participant's degree of mobility and functional ability represented as mean of 10 questions [8 of which relate to participant's functional anatomy and 2 relate to participant's ability to cope with everyday life): 0=easy, 10=impossible; and bath ankylosing spondylitis disease activity index (BASDAI, self-assessment survey of 6 questions for participant's disability due to AS): 0=none, 10=very severe).
Time Frame: Week 14
Population: The intent to treat (ITT) analysis set included all participants who were enrolled and received at least one dose of the study drug and had completed Week 14 visit. Here, N (number of participants analyzed) is defined as the number of participants evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Golimumab (Simponi)
Number analyzed (Participants) | 47
percentage of participants | 74.5

4. Secondary Outcome: Percentage of Psoriatic Arthritis (PsA) Participants Meeting the American College of Rheumatology 20% Improvement Criteria (ACR20) at Week 14
Description: ACR20 was is defined as greater than or equal to (>=) 20% improvement in swollen and tender joint count and >=20% improvement in 3 of following 5 assessments: patient's assessment of pain using Visual Analog Scale (VAS; 0-10 centimeter [cm], 0 cm=no pain and 10 cm=worst possible pain), PGA of disease activity by using VAS (the scale ranges from 0 cm to 10 cm, [0 cm=no pain to 10 cm=worst possible pain]), physician's global assessment of disease activity using VAS (scale ranges from 0 cm to 10 cm; [0 cm=very well and 10 cm=very poor]), participant's assessment of physical function measured by Health Assessment Questionnaire-Disability Index (HAQ-DI, defined as a 20-question instrument assessing 8 functional areas. The derived HAQ-DI ranges from 0, indicating no difficulty, to 3, indicating inability to perform a task in that area) and erythrocyte sedimentation rate (ESR) or C-reactive protein (CRP) level.
Time Frame: Week 14
Population: The ITT analysis set included all participants who were enrolled and received at least one dose of the study drug and had completed Week 14 visit. Here, N (number of participants analyzed) is defined as the number of participants evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Golimumab (Simponi)
Number analyzed (Participants) | 39
percentage of participants | 84.6

5. Secondary Outcome: Percentage of AS Participants With ASAS20 Criteria at Week 24
Description: ASAS 20 response criteria was defined as an improvement from baseline of greater than (>) 20% and >1 unit in at least 3 of following 4 ASAS domains on scale of 0 to 10 units and no worsening from baseline of >20% and >1 unit in the remaining ASAS domain on a scale of 0 to 10 units. The 4 ASAS domains were as follows (0 to 10 units NRS): PGA of disease:0=not active spondylitis, 10=very active spondylitis; total and night Spinal pain: 0=no pain, 10=most severe pain; BASFI, self-assessment of participant's degree of mobility and functional ability represented as mean of 10 questions [8 of which relate to participant's functional anatomy and 2 relate to participant's ability to cope with everyday life): 0=easy, 10=impossible; and BASDAI, self-assessment survey of 6 questions for participant's disability due to AS): 0=none, 10=very severe).
Time Frame: Week 24
Population: The ITT analysis set included all participants who were enrolled and received at least one dose of the study drug and had completed Week 24 visit. Here, N (number of participants analyzed) is defined as the number of participants evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Golimumab (Simponi)
Number analyzed (Participants) | 47
percentage of participants | 66.0

6. Secondary Outcome: Percentage of PsA Participants Meeting the ACR20 Criteria at Week 24
Description: ACR20 was is defined as >=20% improvement in swollen and tender joint count and >=20% improvement in 3 of following 5 assessments: patient's assessment of pain using Visual Analog Scale (VAS; 0-10 centimeter [cm], 0 cm=no pain and 10 cm=worst possible pain), patient's global assessment of disease activity by using VAS (the scale ranges from 0 cm to 10 cm, [0 cm=no pain to 10 cm=worst possible pain]), PGA of disease activity using VAS (scale ranges from 0 cm to 10 cm; [0=very well and 10 cm=very poor]), participant's assessment of physical function measured by HAQ-DI, defined as a 20-question instrument assessing 8 functional areas. The derived HAQ-DI ranges from 0, indicating no difficulty, to 3, indicating inability to perform a task in that area) and ESR or CRP level.
Time Frame: Week 24
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Golimumab (Simponi)
Number analyzed (Participants) | 44
percentage of participants | 93.2

ADVERSE EVENTS:
Time Frame: Up to Week 32
Description: Safety analysis set (SAS) included all participants who were enrolled and received at least one dose of the study intervention.
Arm/Group | Golimumab (Simponi)
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 4/100
Other Adverse Events (participants affected / at risk) | 28/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Golimumab (Simponi) (N=100)
Abdominal Pain (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Irritable Bowel Syndrome (Gastrointestinal disorders) | 1
Lower Respiratory Tract Infection Bacterial (Infections and infestations) | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Golimumab (Simponi) (N=100)
Leukopenia (Blood and lymphatic system disorders) | 1
Vision Blurred (Eye disorders) | 1
Aphthous Ulcer (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Food Poisoning (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 2
Haemorrhoids (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Chills (General disorders) | 1
Pain (General disorders) | 1
Peripheral Swelling (General disorders) | 1
Pyrexia (General disorders) | 4
Body Tinea (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Fungal Infection (Infections and infestations) | 1
Fungal Skin Infection (Infections and infestations) | 1
Herpes Zoster (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 5
Tinea Pedis (Infections and infestations) | 1
Upper Respiratory Tract Infection (Infections and infestations) | 4
Arthropod Sting (Injury, poisoning and procedural complications) | 1
Skin Abrasion (Injury, poisoning and procedural complications) | 1
Blood Bilirubin Increased (Investigations) | 1
Transaminases Increased (Investigations) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 2
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1
Burning Sensation (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Vaginal Discharge (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash Pruritic (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2018-07-02): https://cdn.clinicaltrials.gov/large-docs/25/NCT03733925/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-21): https://cdn.clinicaltrials.gov/large-docs/25/NCT03733925/SAP_001.pdf